CLINICAL TRIAL: NCT03336255
Title: Community Translation of the South Asian Healthy Lifestyle Intervention
Brief Title: South Asian Healthy Lifestyle Initiative (SAHELI)
Acronym: SAHELI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Metropolitan Asian Family Services (Unknown); Skokie Health Department (Unknown); Endeavor Health (Other); Case Western Reserve University (Other); Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Namratha Kandula, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00204939
Record Dates: First submitted 2017-10-19; First posted 2017-11-08 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Print Health Education (No Intervention): Participants will receive primary care referrals and print health education material about heart disease prevention in the mail.
- SAHELI Intervention (Experimental): Participants will enroll in heart disease prevention group sessions focusing on physical activity, diet, weight, and stress management. Each group will have 16 to 20 participants who will attend 16 weekly, 90 minute group education sessions at Metropolitan Asian Family Services or Skokie Health Department. During each session, participants will watch videos on the day's topic followed by discussion, activities, and assistance in setting realistic goals with attention to physical activity, diet, weight, and stress management.
  Interventions: Behavioral: South Asian Healthy Lifestyle Initiative (SAHELI)

INTERVENTIONS:
Behavioral: South Asian Healthy Lifestyle Initiative (SAHELI) — Culturally tailored lifestyle intervention for South Asians.
  Other Names: SAHELI
  Arms: SAHELI Intervention

SUMMARY:
Research show that South Asians (SA) have a high burden of Cardiovascular Disease (CVD) risk factors of which, poor diet and physical inactivity remain the major lifestyle risk factors in SA. Intensive diet and physical activity behavioral interventions have been shown to yield improvements across a variety of intermediate cardiovascular health outcomes (blood pressure, cholesterol, glycated hemoglobin, weight) in persons with CVD risk factors and are recommended by national guidelines. However, the investigators prior research found that existing interventions are not reaching SA. First, the usual framing of behavioral risk factor interventions in terms of the biomedical model of CVD is mismatched to SA explanatory models, which emphasize psychosocial causes of CVD. Next, few interventions are tailored to the sociocultural patterns shared by much of the SA community. Interventions that address the individual and shared sociocultural drivers of CVD risk are needed to maximize reach and effectiveness in the high risk and rapidly growing SA population. The proposed study builds on the strong foundation of the South Asian Healthy Lifestyle Initiative (SAHELI), which has a 9-year history of using community-based participatory research to design and test culturally tailored, community-based interventions to reduce CVD disparities in SA. To date, SAHELI has engaged multi-sectoral partners, established relationships of trust, and defined mutually beneficial goals. The investigators also culturally adapted the SAHELI lifestyle intervention to (a) address the individual and sociocultural determinants of CVD risk in SA; and (b) increase components of self-regulation (motivation, self-monitoring, goal setting) that are most effective in eliciting diet and physical activity changes. Hence, the SAHELI intervention integrates evidence-based behavior change techniques with the shared the sociocultural processes salient to SA. A pilot study (n=63) established feasibility of the SAHELI intervention, had a 100% retention rate, and reduced glycated hemoglobin and weight among intervention participants compared to a control group. The proposed study is based on the pilot study and will use a hybrid trial type 1 design to evaluate the clinical effectiveness and implementation potential of the culturally tailored, community-based lifestyle intervention in a larger, more generalizable at-risk SA population. Study team is uniquely positioned to fill a critical gap in work (a) demonstrating the cultural adaptation of evidence-based lifestyle interventions, and (b) evaluating the effectiveness of the SAHELI intervention in reducing CVD risk in SA living in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* South Asian adults (18-65 years)
* Living within the 22 square mile study area
* Ability to understand Hindi, Urdu, Gujarati or English. AND

Body Mass Index of 25 and over and a diagnosis by a doctor of high cholesterol or pre-diabetes/Diabetes, or High blood pressure. OR Body Mass Index of 23 to 24.9 and one clinical risk factors for Cardiovascular Disease (CVD) (CVD risk factors are: Hypertension (Systolic blood pressure >=130 or diastolic blood pressure >=80), abnormal cholesterol (Total cholesterol ≥200, triglycerides >=150),pre-diabetes (A1c between 5.7-6.4%), or diabetes (A1c 6.5 to 10.9),

Exclusion Criteria:

* History of a CVD event (stroke or heart attack)
* Being on insulin
* Blood pressure ≥180/100 mmHg
* HbA1c ≥11% BMI ≥ 40
* Current pregnancy
* Being ≤ 12 months postpartum
* Any underlying diseases likely to limit lifespan and/or affects ability to exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2023-02-11 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Participants who receive SAHELI intervention may show greater reduction in clinical risk factors for cardiovascular disease compared to the control group. | 12 months
  Total of 550 participants with 50% randomized to SAHELI intervention arm will show significantly greater improvements in clinical risk factors associated with Cardio Vascular Disease (primary outcomes of systolic and diastolic blood pressure, cholesterol, glycated hemoglobin, and weight) relative to a comparison group that receives print education materials on healthy lifestyle.

CONTACTS AND LOCATIONS:
Overall Officials: Namratha Kandula, MD,MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kandula NR, Bernard V, Dave S, Ehrlich-Jones L, Counard C, Shah N, Kumar S, Rao G, Ackermann R, Spring B, Siddique J. The South Asian Healthy Lifestyle Intervention (SAHELI) trial: Protocol for a mixed-methods, hybrid effectiveness implementation trial for reducing cardiovascular risk in South Asians in the United States. Contemp Clin Trials. 2020 May;92:105995. doi: 10.1016/j.cct.2020.105995. Epub 2020 Mar 24. PMID 32220632
- [Result] Lam EL, Kandula NR, Shah NS. The Role of Family Social Networks in Cardiovascular Health Behaviors Among Asian Americans, Native Hawaiians, and Pacific Islanders. J Racial Ethn Health Disparities. 2023 Oct;10(5):2588-2599. doi: 10.1007/s40615-022-01438-9. Epub 2022 Nov 3. PMID 36329308
- [Result] Vu M, Nedunchezhian S, Lancki N, Spring B, Brown CH, Kandula NR. A mixed-methods, theory-driven assessment of the sustainability of a multi-sectoral preventive intervention for South Asian Americans at risk for cardiovascular disease. Implement Sci Commun. 2024 Sep 13;5(1):89. doi: 10.1186/s43058-024-00626-4. PMID 39267181
- [Result] Kandula NR, Shah NS, Kumar S, Charley M, Clauson M, Lancki N, Finch EA, Ehrlich-Jones L, Rao G, Spring B, Shah NS, Siddique J. Culturally Adapted Lifestyle Intervention for South Asian Adults With Cardiovascular Risk Factors: The SAHELI Randomized Clinical Trial. JAMA Cardiol. 2024 Nov 1;9(11):973-981. doi: 10.1001/jamacardio.2024.2526. PMID 39259546